CLINICAL TRIAL: NCT00643383
Title: A Two-Arm Study Comparing the Analgesic Efficacy and Safety of Acetaminophen and Tramadol Combination BID Versus Placebo for the Treatment of Acute Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06CCL3-001; NCT00643383 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Acute Low Back Pain
MeSH Terms: interventions — Drug Combinations; Acetaminophen; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Combination drug (Acetaminophen + Tramadol)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Combination drug (Acetaminophen + Tramadol)
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
A multi-center placebo controlled, double-blind, trial comparing the analgesic efficacy and safety of Acetram Contramid® BID versus placebo for the treatment of acute low back pain in patients between 18 and 80 yrs of age.

ELIGIBILITY:
Inclusion Criteria:

* Males or females in generally good health aged 18-80 years with moderate to severe acute low back pain.
* Current acute low back pain episode within 48h prior to study entry.
* Pain must be moderate to severe following incident

Exclusion Criteria:

* Chronic low back pain
* Ongoing or history of alcohol or drug abuse
* Body Mass Index greater 39
* Treatment within the last 3 weeks with monoamine oxidase inhibitors; tricyclic antidepressants and other tricyclic compounds; neuroleptics; selective serotonin reuptake inhibitors
* Known history or symptoms suspicious for cancer
* Significant renal or liver disease
* Spinal surgery within 1 year of study entry.
* Subjects who are pregnant or lactating.
* Subjects with unstable medical disease.
* Subjects who have received treatment with an investigational product/device with 30 days prior to study entry.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Pain Intensity change from Baseline

SECONDARY OUTCOMES:
Overall satisfaction with the study medication
Safety evaluation

CONTACTS AND LOCATIONS:
Locations (33):
- United States (17):
  - Montgomery, Alabama
  - Centennial, Colorado
  - Hialeah, Florida
  - Largo, Florida
  - New Port Richey, Florida
  - Indianapolis, Indiana
  - Waterloo, Iowa
  - Baton Rouge, Louisiana
  - Brockton, Massachusetts
  - Minneapolis, Minnesota
  - Oklahoma City, Oklahoma
  - Rapid City, South Dakota
  - Crossville, Tennessee
  - Bryan, Texas
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
- Canada (16):
  - Bathurst, New Brunswick
  - Mount Pearl, Newfoundland and Labrador
  - Greater Sudbury, Ontario
  - Newmarket, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Cowansville, Quebec
  - Drummondville, Quebec
  - Gatineau, Quebec
  - Granby, Quebec
  - Mirabel, Quebec
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
  - Trois-Rivières, Quebec

REFERENCES:
- [Derived] Lasko B, Levitt RJ, Rainsford KD, Bouchard S, Rozova A, Robertson S. Extended-release tramadol/paracetamol in moderate-to-severe pain: a randomized, placebo-controlled study in patients with acute low back pain. Curr Med Res Opin. 2012 May;28(5):847-57. doi: 10.1185/03007995.2012.681035. Epub 2012 Apr 25. PMID 22458917